CLINICAL TRIAL: NCT05189756
Title: Dual-dose Aprepitant to Reduce Postoperative Nausea and Vomiting After Laparoscopic Bariatric Surgery: a Prospective, Randomised, Placebo-controlled, Triple-blind, Single Centre Trial.
Brief Title: Dual-dose Aprepitant to Reduce Postoperative Nausea and Vomiting After Laparoscopic Bariatric Surgery.
Acronym: DDA-PONV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruiting rate
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BECD-2-21
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Nausea and Vomiting; Bariatric Surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomised, placebo-controlled, triple-blind, single centre, two-arm parallel groups superiority trial assessing incidence of PONV 48 hours after laparoscopic bariatric surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Verum, placebo and block-randomisation will be provided by hospital pharmacy. Therefore, patients, treating team and researcher will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum (Experimental): Patients will receive 2 encapsulated capsules containing aprepitant 80mg to be ingested with a sip of water 2 hours before surgery and 24 hours after surgery. Surgery will follow our hospital enhanced recovery after surgery (ERAS) standard (general anaesthesia using volatile anaesthetics, intravenous dexamethasone 8mg and ondansetron 4mg for PONV prophylaxis).
  Interventions: Drug: Aprepitant 80 mg
- Placebo (Placebo Comparator): Patients will receive similar looking encapsulated capsules containing only placebo to be ingested with a sip of water 2 hours before surgery and 24 hours after surgery. Surgical and anaesthetic procedures are identical to the verum arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprepitant 80 mg — Encapsulated capsule of aprepitant 80mg to make it look alike to the placebo.
  Other Names: Aprepitant Zentiva 80mg
  Arms: Verum
Drug: Placebo — Encapsulated placebo capsules for optical, acoustical and haptic blinding.
  Other Names: Placebo Capsules
  Arms: Placebo

SUMMARY:
Postoperative nausea and vomiting (PONV) is unpleasant and increases health care costs. Despite modern techniques and prophylaxis, PONV rates remain high after laparoscopic bariatric surgery. We aim to reduce PONV after laparoscopic bariatric surgery using aprepitant with a similar scheme used for emetogenic chemotherapy.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is not only a disturbing and unpleasant experience for the patient, it also increases length of post anaesthesia care unit (PACU) and hospital stay. In addition, PONV increases the risk for unplanned admission, risk for complications and in the end, health care costs. Risk factors have been identified more than 20 years ago by Apfel et. al., whose screening score has been widely implemented to augment perioperative prophylaxis. But despite modern anaesthetic techniques and combined antiemetic prophylaxis, PONV rates remain high in patients at high risk for PONV: in a recent retrospective study in female patients after laparoscopic bariatric surgery, up to 68% suffered from PONV during the first 48 hours after surgery despite triple antiemetic prophylaxis. While aprepitant is prescribed for three consecutive days after chemotherapy, there is no study so far evaluating the effect of a second dose of aprepitant 24 hours after surgery to prevent the increase in PONV after PACU discharge. We hypothesise, that adding two scheduled doses of aprepitant (2 hours before and 24 hours after surgery) to a twofold antiemetic regimen will significantly reduce cumulative PONV in the first 48 hours after laparoscopic bariatric surgery in patients with moderate to high risk for PONV.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and more
* Scheduled for an elective, laparoscopic bariatric surgery (either laparoscopic gastric sleeve resection or laparoscopic gastric bypass)
* BMI > 30 kg/m2
* moderate to high risk for PONV (defined as APFEL score of 2 or higher)
* Informed Consent as documented by signature (see appendix 2).

Exclusion Criteria:

* emergency or open abdominal surgery;
* contraindication to aprepitant:

  * known allergy/hypersensitivity
  * on pimozide, terfenadine, astemizole or cisapride
* on regular medication with known interaction with the study drug:

  * benzodiazepines
  * ketoconazole, itraconazole
  * rifampicin, clarithromycin
  * paroxetine
  * diltiazem
  * carbamazepine, phenytoin
  * tolbutamid
  * ritonavir
  * St. John's wort
* patients with history of chronic nausea/vomiting or taking medication with known antiemetic properties (dexamethasone, metoclopramide, meclozine)
* severe hepatic impairment (Child-Pugh score >9);
* chronic substance abuse (except smoking);
* significant psychiatric disease precluding interrogation;
* Inability to follow the procedures of the study, e. g. due to language barrier;
* Women who are pregnant or breast feeding;
* Intention to become pregnant during the course of the study and 2 months after surgery;
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a condom in addition to a medically reliable method of contraception for the entire study duration and 2 months after surgery, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* male participants need to use a condom for the whole study period and 2 months after surgery;
* unable to consent, e. g. patients incapable of judgment needing next-of-kin consent or under tutelage;
* participation in another study with an investigational drug within the 30 days preceding and during the present study;
* previous enrolment into the current study;
* enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Cumulative rate of PONV 48 hours after surgery | 48 hours
  Primary outcome is cumulative rate of PONV (defined as emesis including vomiting and retching, severe nausea [>6/10 on a numeric rating scale (NRS)] and use of rescue medication) at 48 hours after surgery.

SECONDARY OUTCOMES:
Severity of nausea | 3, 24 and 48 hours after surgery
  mild [NRS 1-3], moderate [NRS 4-6] and severe [NRS 7-10]
Incidence of emesis | 3, 24 and 48 hours after surgery
  number
Use of rescue medication for PONV | 3, 24 and 48 hours after surgery
  medication, cumulative dose, route
Use of opioid analgesics | 3, 24 and 48 hours after surgery
  mg of oral morphine equivalents
Use of non-opioid analgesics | 3, 24 and 48 hours after surgery
  medication, cumulative dose, route
Use of co-analgesics | 3, 24 and 48 hours after surgery
  medication, cumulative dose, route
Rate of delayed PACU discharge because of PONV | 24 hours after surgery
  number
Length of PACU stay | 24 hours after surgery
  hours
Length of hospital stay | 48 hours after surgery
  hours
Surgical complications at 30 days after surgery | 30 days
  using Clavien-Dindo classification (number and grade)

OTHER OUTCOMES:
Adverse Events | 3, 24 and 48 hours after surgery, 30 days after surgery
  pre-defined events, safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Christian M Beilstein, MD, Principal Investigator — Bern University Hospital, University of Bern, Bern, Switzerland
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Bern University Hospital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No